CLINICAL TRIAL: NCT01186042
Title: Chronic HIV Infection and Aging in NeuroAIDS (CHAIN)
Acronym: CHAIN
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0396-10-FB; P30MH062261 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-08-20 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: HIV; Aging
Keywords: HIV; Aging; Neuropsychological function; Activity; Sleep patterns; Frailty; Emotional well-being; Sexual health
MeSH Terms: conditions — Motor Activity; Frailty | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aging in HIV: 20-40 years of age or older than 50
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention

SUMMARY:
The purpose of this study is to find the best tests to use to investigate the differences between older and younger people with HIV disease. Test to be included will measures of memory, learning, activity levels, sleep patterns, emotional well-being and sexual health.

DETAILED DESCRIPTION:
Advances in the treatment of chronic HIV disease over the last 20 years have resulted in dramatic declines in morbidity and mortality. However, emerging data suggest that chronically infected patients may be aging prematurely, and/or experience increased incidence of age-related conditions. These phenomena are poorly understood. The overall goal of the CHAIN project is to support the expansion of innovative research on the effects of chronic HIV infection, co-morbidities, and aging on the central nervous system (CNS). We propose the initiation of a clinical portion to better understand the nature of the aging process in HIV-infected patients, with an emphasis on brain disease. This is a pilot, feasibility study to inform the design of a larger, prospective cohort study.

We plan to enroll 20 older HIV-infected patients (more than 50 years old) and 20 younger controls (20-40 years old), matched for gender and race/ethnicity. Participants will undergo a series of tests, at one comprehensive assessment. Demographic and medical history data will be abstracted from the medical record. Each participant will undergo a medical history and physical examination, and a battery of tests designed to evaluate neuropsychological function, activity, sleep patterns, frailty, emotional well-being and sexual health. These will consist of self-administered questionnaires and neuropsychological tests, as detailed in the Methods section. Innovative measures will be included such as an activity monitor worn by participants, and a Wii balance board to assess standing balance. Participants will be asked to keep a diary and wear the activity monitoring device for one month. Plasma and serum samples will be collected on one occasion for future testing of potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV infection.
* 20-40 years of age or older than 50.
* If taking antiretroviral therapy, on stable therapy for the past 12 weeks and not anticipated to require a change in therapy during the following 6 weeks.
* If not taking antiretroviral therapy, not anticipated to initiate therapy in the next 6 weeks.
* Ability to provide written informed consent.
* Ability to complete the questionnaires in English.

Exclusion Criteria:

* Completion of treatment for any intercurrent acute infection less than four weeks before study entry. Maintenance or prophylactic therapy is permitted for opportunistic infections.
* Any active psychiatric illness including schizophrenia, severe depression, or severe bipolar affective disorder that, in the opinion of the investigator, could confound performance of or the analysis of the test results.
* Active drug or alcohol abuse that, in the investigator's opinion, could compromise compliance with study procedures or confound the analysis of the test results.
* Major neurologic disease such as multiple sclerosis or stroke, active brain infection (except for HIV-1), brain neoplasm, or space-occupying brain lesion.
* Current delirium or intoxication.
* Pregnancy.
* Any other condition that, in the opinion of the investigator, is a contraindication to participation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Nebraska Medical Center HIV Clinic
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of enrolling older HIV-infected patients and younger controls into a prospective, observational study. | One month
  Evaluate the feasibility of enrolling older HIV-infected patients and youger controls into a prospective, observational study.

SECONDARY OUTCOMES:
Selection of the optimal test battery to measure the areas of interest | One month
  Secondary objective includes:
  Selection of the optimal test battery to measure the areas of interest;
Participant acceptance of the measures involved | One month
  Secondary objective includes:
  Participant acceptance of the measures involved;
Preliminary data collection to inform the size and design of a larger, follow-up study. | One month
  Secondary objective includes:
  Preliminary data collection to inform the size and design of a larger, follow-up study.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Swindells, MBBS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Valcour V, Shikuma C, Shiramizu B, Watters M, Poff P, Selnes O, Holck P, Grove J, Sacktor N. Higher frequency of dementia in older HIV-1 individuals: the Hawaii Aging with HIV-1 Cohort. Neurology. 2004 Sep 14;63(5):822-7. doi: 10.1212/01.wnl.0000134665.58343.8d. PMID 15365130
- See also: University of Nebraska Medical Center HIV Clinic — http://www.unmc.edu/hiv